CLINICAL TRIAL: NCT00378287
Title: A Randomized, Controlled, Double-blind, Cross-over Study of the Effect of Oral Rabeprazole 20mg and Intravenous Pantoprazole 40mg on Intragastric pH in Patients
Brief Title: A Study to Monitor Intragastric pH in Patients Taking Rabeprazole vs. Patients Taking Pantoprazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR005824
Record Dates: First submitted 2006-09-15; First posted 2006-09-19 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: GERD
Keywords: Acid Reflux; Proton Pump Inhibitor; GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

INTERVENTIONS:
Drug: rabeprazole sodium

SUMMARY:
The purpose of the study is to demonstrate in patients that oral rabeprazole produces equivalent acid suppression to intravenous pantoprazole on Day 1 of drug administration.

DETAILED DESCRIPTION:
Following screening to determine eligibility (normal medical history, physical examination including vital signs, laboratory findings, negative test for active H. pylori infection, and a negative pregnancy test if applicable) and subsequent enrolment, patients will have a baseline 24-hour intragastric pH recording. Patients will receive either oral rabeprazole 20mg or intravenous pantoprazole 40mg daily for 3 consecutive days. For blinding purposes, patients will also receive either a placebo oral tablet or placebo intravenous solution ("double-dummy" design). A 24-hour intragastric pH recording will be completed on Day 1 and Day 3 of the drug administration period. This will be followed by a 14-day washout period before the second 3-day drug administration period during which the patient will receive the crossover drug regimen, and will again have 24-hour intragastric pH recordings completed on the first and third days of this second drug administration period.Thirty-seven patients with a negative test for active H. pylori infection test will be randomised into the study. The primary hypothesis is that oral rabeprazole produces equivalent acid suppression to intravenous pantoprazole as indicated by the time during which intragastric pH is greater than 4 on Day 1 of drug administration. Eligible patients will be randomly assigned to 1 of the 2 treatment groups and will first receive either oral rabeprazole 20mg plus placebo intravenous solution or intravenous pantoprazole 40mg plus a placebo oral tablet daily for 3 consecutive days. After a 14-day washout, patients will receive the crossover drug regimen.

Rabeprazole: supplied as 20mg tablets (and matching placebo tablets). Pantoprazole: supplied as 12-mL vials of lyophilized powder containing pantoprazole 40mg (pantoprazole

ELIGIBILITY:
Inclusion Criteria:

* Female patients must be postmenopausal (for at least 1 year), sterile (6 months post-sterilization), or practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study. Patients of childbearing potential (including those using birth control) must have a negative pregnancy serum test at screening before medication is dispensed
* Absence of Hp infection, as established by a negative 13C-urea breath test (13C-UBT)
* Body mass index (BMI) between 18-33 kg/m2, and weight between 50 and 135kg. BMI calculation: BMI = weight (kg) / height (m) 2

Exclusion Criteria:

* Documentation of significant past history of gastrointestinal disease requiring therapy
* Patients with a baseline pH recording indicative of an abnormal acid secretory pattern
* Significant concurrent disease or clinical illness within 14 days of initial screening visit
* Use of any prescription medications within 14 days of initial screening visit, with the exception of oral contraceptive medications, and non-systemic medications such as topical medications for skin conditions, or nasal sprays for allergy relief
* Use of either over-the-counter (OTC) or prescription histamine-2 receptor antagonists (H2RAs), and/or proton pump inhibitors (PPIs) prokinetics, antibiotics or bismuth compounds within 28 days of the screening 13C-UBT
* Use of any OTC medication within 7 days of the initial screening visit, with the exception of acetaminophen (up to a daily maximum of 2g), and OTC eye drops, nasal drops or sprays for allergy relief.10.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-10; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is the percentage of time intragastric pH >4 for the 24-hour monitoring period on Day 1 (i.e.: first day of dosing for each treatment period).

SECONDARY OUTCOMES:
Percentage of time intragastric pH is >3, >4, >5, >6 on Day 1, and on Day 3 over time intervals: 0-14h and 14-24h after dosing;Median intragastric pH on Day 1 and Day 3 (entire 24-hour interval, and over time intervals: 0-14h and 14-24h after dosing)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada

REFERENCES:
- [Result] Armstrong D, James C, Camacho F, Chen Y, Horbay GL, Teixeira B, Husein-Bhabha FA. Oral rabeprazole vs. intravenous pantoprazole: a comparison of the effect on intragastric pH in healthy subjects. Aliment Pharmacol Ther. 2007 Jan 15;25(2):185-96. doi: 10.1111/j.1365-2036.2006.03160.x. Epub 2006 Nov 16. PMID 17116123
- See also: A Randomized, Controlled, Double-blind, Cross-over Study of the Effect of Oral Rabeprazole 20mg and Intravenous Pantoprazole 40mg on Intragastric pH in Patients — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=362&filename=CR005824_CSR.pdf